CLINICAL TRIAL: NCT00424957
Title: Brain Energy Metabolism in Patients With Acute Hepatic Encephalopathy Measured With PET
Brief Title: Brain Energy Metabolism in Patients With Chronic Liver Disease and Impaired Central Nervous System
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Peter Iversen, PET Center, Aarhus University Hospital
Other Study IDs: 20060120
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Cirrhosis; Hepatic Encephalopathy
Keywords: Ammonia; Astrocytes; Citric acid cycle; Alpha ketoglutarate dehydrogenase
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the current study is to look into the pathogenesis of a severe medical condition causing acute episodes on the central nervous system as seen in majority of patients with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* 6 patients with liver cirrhosis with an acute episode of hepatic encephalopathy,
* 6 patients with liver cirrhosis without an acute episode of hepatic encephalopathy,
* 6 healthy subjects age and sex matched

Exclusion Criteria:

* Neurological and/or psychiatric condition,
* Non-treated diabetes,
* Pregnancy/breast-feeding

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 6 patients with liver cirrhosis with an acute episode of hepatic encephalopathy, 6 patients with liver cirrhosis without an acute episode of hepatic encephalopathy, 6 healthy subjects age and sex matched
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Keiding, MD, Study Chair — PET Centre and Medical department V, Aarhus Sygehus, Aarhus University Hospital
Locations (1):
- PET Centre, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Ott P, Clemmesen O, Larsen FS. Cerebral metabolic disturbances in the brain during acute liver failure: from hyperammonemia to energy failure and proteolysis. Neurochem Int. 2005 Jul;47(1-2):13-8. doi: 10.1016/j.neuint.2005.04.002. PMID 15921824